CLINICAL TRIAL: NCT00540124
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Pilot Study to Evaluate the Efficacy and Safety of Tadalafil and Tamsulosin Once-a-Day Dosing for 12 Weeks in Asian Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: Pilot Study Investigating Safety and Efficacy of Tadalafil as Treatment for Benign Prostatic Hyperplasia (BPH) in Asian Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11658; H6D-MC-LVHT (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Results first posted 2009-07-20 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tadalafil (Experimental)
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Tamsulosin (Active Comparator)
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tadalafil — 5 mg once a day
  Other Names: LY450190; Cialis
  Arms: Tadalafil
Drug: Placebo — once a day
  Arms: Placebo
Drug: Tamsulosin — 0.2 mg once a day
  Arms: Tamsulosin

SUMMARY:
The primary purpose of this clinical trial is to evaluate the change in the International Prostate Symptom Score (IPSS) total score from the beginning of the study to the end of the study for subjects randomized to tadalafil 5mg once a day dosing and placebo once a day dosing for 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have Benign Prostatic Hyperplasia - Lower Urinary Tract Symptoms (BPH-LUTS) for at least 6 months prior to Visit 1.
* Agree not to use any other approved or experimental treatments for erectile dysfunction or BPH-LUTS during the study.
* Have not taken Finasteride therapy for at least 3 months prior to Visit 2.
* Have not taken Dutasteride therapy for at least 6 months prior to Visit 2.
* Have an International Prostate Symptom Score (IPSS) total score greater than or equal to 13 at Visit 2.

Exclusion Criteria:

* Prostate Specific Antigen (PSA) greater than 10.0 nanograms per milliliter (ng/mL) at Visit 1.
* Bladder Post Void Residual (PVR) greater than or equal to 300 mL by ultrasound at Visit 1.
* History of pelvic surgery, prostatectomy, radiotherapy, penile implant surgery, lower urinary tract malignancy or trauma.
* Urinary tract infection or inflammation or current antibiotic therapy for urinary tract infection at Visit 1.
* Glycosylated hemoglobin (HbA1c) greater than 9% at Visit 1.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- South Korea (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeonju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyunggi-Do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pusan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were three periods to this study. Period 1 was a 4-week Screening/Washout Period. 196 subjects screened (45 failures). Period 2 was a 4-week Placebo Run-in Period. Period 3 was a 12-week Treatment Period (151 subjects randomized).
Groups:
- Placebo: by mouth once a day
- Tadalafil: 5 mg by mouth once a day
- Tamsulosin: 0.2 mg by mouth once a day
Period: Overall Study
Arm/Group | Placebo | Tadalafil | Tamsulosin
Started | 51 | 51 | 49
Completed | 47 | 48 | 48
Not Completed | 4 | 3 | 1
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Entry Criteria Not Met | 2 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Tamsulosin | Total
Number analyzed (Participants) | 51 | 51 | 49 | 151
Age Continuous [Mean (Standard Deviation); unit: years] | 62.2 (6.8) | 61.2 (6.6) | 61.5 (6.4) | 61.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 51 | 51 | 49 | 151
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 51 | 51 | 49 | 151
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 51 | 51 | 49 | 151
Erectile Dysfunction (ED) [Number; unit: participants]
  Yes | 36 | 30 | 24 | 90
  No | 15 | 21 | 25 | 61
Duration of Erectile Dysfunction (ED) [Number; unit: participants] — Because this measure applies only to participants with ED, the number of participants reported here will be less than the total number of participants in the study.
  participants
    <3 Months | 0 | 1 | 0 | 1
    3 Months to < 6 Months | 2 | 3 | 1 | 6
    6 Months to < 1 Year | 5 | 3 | 5 | 13
    1 Year or More | 29 | 23 | 18 | 70
Etiology of Erectile Dysfunction (ED) [Number; unit: participants] — Because this measure applies only to participants with ED, the number of participants reported here will be less than the total number of participants in the study.
  participants
    Psychogenic | 2 | 0 | 0 | 2
    Organic | 16 | 10 | 11 | 37
    Mixed | 17 | 15 | 12 | 44
    Unknown | 1 | 5 | 1 | 7
Severity of Erectile Dysfunction (ED) [Number; unit: participants] — Because this measure applies only to participants with ED, the number of participants reported here will be less than the total number of participants in the study. Severity is determined from the International Index of Erectile Function Scores. Scores range from 0 (low or no erectile function) to 5 (high erectile function) on 6 questions (1-5, 15 of the IIEF). Total Erectile Function Domain scores range from 0 to 30. Severity is determined based on scores as follows:
  Severe ED ≤10 Moderate ED 11-16 Mild ED 17-25 No ED >25
  participants
    Mild | 17 | 22 | 13 | 52
    Moderate | 14 | 5 | 7 | 26
    Severe | 5 | 3 | 4 | 12
Lower Urinary Tract Symptoms Severity [Number; unit: participants] — Severity was assessed through the International Prostate Symptom (IPSS) Total Score. The Total Score was obtained by combining the scores of the responses to 1 through 7 component questions. Each question is scored from 0-5 for a range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
  participants
    Moderate (IPSS < 20) | 35 | 35 | 33 | 103
    Severe (IPSS ≥20) | 16 | 16 | 16 | 48
Postvoid Residual Volume (PRV) [Mean (Standard Deviation); unit: milliliters] | 34.4 (35.7) | 30.9 (33.8) | 42.0 (59.6) | 35.7 (44.3)
Height [Mean (Standard Deviation); unit: centimeters] | 168.6 (5.2) | 168.6 (5.5) | 167.3 (4.6) | 168.2 (5.1)
Weight [Mean (Standard Deviation); unit: kilograms] | 70.7 (8.1) | 70.1 (7.5) | 68.4 (7.6) | 69.7 (7.7)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meters squared (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/meters squared (kg/m^2) | 24.8 (2.2) | 24.7 (2.3) | 24.4 (2.1) | 24.6 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Week Endpoint in International Prostate Symptom Score (IPSS) Total Score
Description: The IPSS Total Score is obtained by combining the scores of the responses to 1 through 7 component questions. Each question is scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: baseline, 12 weeks
Population: Primary analysis was performed on an intent-to-treat basis. Data from participants with baseline and at least one post-baseline data were used for the analysis. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 50 | 50 | 49
units on a scale
  Baseline | 17.3 (5.0) | 17.1 (5.4) | 17.7 (5.0)
  12 Week Change | -4.2 (4.8) | -5.8 (4.6) | -5.6 (5.3)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.073, ANCOVA — P-value for 12 Week Change. Change=Endpoint minus baseline. P-values are from an ANCOVA with effects for treatment, prior alpha blocker use (yes/no), and baseline value, and were not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.186, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline to 4 Week and 8 Week Endpoints in International Prostate Symptom Score (IPSS) Total Score
Description: as for outcome 1
Time Frame: baseline, 4 and 8 weeks
Population: Secondary continuous analyses were performed on an intent-to-treat basis. Data from participants with baseline and at least one post-baseline data were used for the analysis. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 50 | 50 | 49
units on a scale
  4 Week Change (n=50, n=49, n=49) | -2.8 (0.6) | -4.0 (0.6) | -4.0 (0.6)
  8 Week Change (n=47, n=50, n=48) | -3.3 (0.7) | -4.8 (0.6) | -4.8 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.155, ANCOVA — P-value for 4 Week Change. Change=Endpoint minus baseline. P-values are from an ANCOVA with effects for treatment, prior alpha blocker use (yes/no), and baseline value, and were not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.155, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.108, ANCOVA — P-value for 8 Week Change. Change=Endpoint minus baseline. P-values are from an ANCOVA with effects for treatment, prior alpha blocker use (yes/no), and baseline value, and were not adjusted for multiple comparisons
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.112, ANCOVA — [p-value comment as in outcome 2, analysis 3]

3. Secondary Outcome: Change From Baseline to 4, 8, and 12 Week Endpoints in International Prostate Symptom Score (IPSS) - Irritative Subscore
Description: The IPSS storage (irritative) subscore is defined as sum of scores for Questions 2, 4, and 7 of the IPSS. If scores for any of these questions are missing for a visit, the IPSS storage subscore will be reported as missing for that visit. Subscore totals range from 0 to 15; higher scores are indicative of greater irritation.
Time Frame: baseline, 4, 8, and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 50 | 50 | 49
units on a scale
  Baseline (n=50, n=50, n=49) | 6.7 (2.0) | 6.7 (2.7) | 6.5 (2.6)
  4 Week Change (n=50, n=49, n=49) | -0.8 (2.1) | -1.4 (2.4) | -1.7 (2.1)
  8 Week Change (n=47, n=50, n=48) | -0.9 (2.0) | -1.6 (2.5) | -1.9 (2.3)
  12 Week Change (n=47, n=48, n=48) | -1.6 (2.1) | -2.2 (2.4) | -1.8 (2.7)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.137, ANCOVA — P-value for 4 Week Change. Change=Endpoint minus baseline. P-values are from ANCOVA with effects for treatment, prior alpha blocker use (yes/no), time (visit), baseline value, and time*treatment interaction. Model used an unstructured covariance
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.009, ANCOVA — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.118, ANCOVA — P-value for 8 Week Change. Change=Endpoint minus baseline. P-values are from ANCOVA with effects for treatment, prior alpha blocker use (yes/no), time (visit), baseline value, and time*treatment interaction. Model used an unstructured covariance
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.018, ANCOVA — [p-value comment as in outcome 3, analysis 3]
Statistical Analysis 5: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.207, ANCOVA — P-value for 12 Week Change. Change=Endpoint minus baseline. P-values are from ANCOVA with effects for treatment, prior alpha blocker use (yes/no), time (visit), baseline value, and time*treatment interaction. Model used an unstructured covariance
Statistical Analysis 6: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.581, ANCOVA — [p-value comment as in outcome 3, analysis 5]

4. Secondary Outcome: Change From Baseline to 4, 8, and 12 Week Endpoints in International Prostate Symptom Score (IPSS) - Obstructive Subscore
Description: The IPSS voiding (obstructive) subscore is defined as sum of scores for Questions 1, 3, 5, and 6 of the IPSS. If scores for any of these questions are missing for a visit, the IPSS voiding subscore will be reported as missing for that visit. Subscore totals range from 0 to 20; higher scores are indicative of greater obstruction.
Time Frame: baseline, 4, 8, and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 50 | 50 | 49
units on a scale
  Baseline (n=50, n=50, n=49) | 10.6 (3.7) | 10.4 (3.8) | 11.2 (3.7)
  4 Week Change (n=50, n=49, n=49) | -2.0 (4.0) | -2.6 (3.1) | -2.4 (3.1)
  8 Week Change (n=47, n=50, n=48) | -2.3 (4.1) | -3.1 (3.1) | -3.1 (3.8)
  12 Week Change (n=47, n=48, n=48) | -2.7 (3.6) | -3.6 (3.4) | -3.9 (3.6)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.306, ANCOVA — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.762, ANCOVA — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.203, ANCOVA — [p-value comment as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.464, ANCOVA — [p-value comment as in outcome 3, analysis 3]
Statistical Analysis 5: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.169, ANCOVA — [p-value comment as in outcome 3, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.243, ANCOVA — [p-value comment as in outcome 3, analysis 5]

5. Secondary Outcome: Change From Baseline to 4, 8, and 12 Week Endpoints in International Prostate Symptom Score (IPSS) - Nocturia Subscore
Description: IPSS Question 7 is used to assess the frequency of nocturia. Scores range from 0 (low frequency of nocturia) to 5 (high frequency of nocturia).
Time Frame: baseline, 4, 8, and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 50 | 50 | 49
units on a scale
  Baseline (n=50, n=50, n=49) | 2.0 (1.1) | 1.8 (1.0) | 1.7 (1.0)
  4 Week Change (n=50, n=49, n=49) | -0.3 (0.9) | -0.4 (0.9) | -0.3 (1.0)
  8 Week Change (n=47, n=50, n=48) | -0.4 (0.7) | -0.4 (1.0) | -0.4 (1.2)
  12 Week Change (n=47, n=48, n=48) | -0.5 (0.9) | -0.5 (0.9) | -0.5 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.206, ANCOVA — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.457, ANCOVA — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.892, ANCOVA — [p-value comment as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.593, ANCOVA — [p-value comment as in outcome 3, analysis 3]
Statistical Analysis 5: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.887, ANCOVA — [p-value comment as in outcome 3, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.762, ANCOVA — [p-value comment as in outcome 3, analysis 5]

6. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Benign Prostatic Hyperplasia Impact Index (BPH-II)
Description: The BPH-BII is a 4-item, self-administered questionnaire evaluating impact of urinary problems on overall health and activity. Total scores range of 0 to 13; higher scores represent increased perceived impact of BPH-LUTS on overall health. If scores for any component question were missing for a visit, BPH-BII was reported as missing for that visit.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 48 | 49 | 48
units on a scale
  Baseline | 6.2 (2.8) | 6.1 (2.9) | 6.2 (3.1)
  12 Week Change | -2.0 (2.7) | -2.2 (2.9) | -1.7 (2.6)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.691, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.415, ANCOVA — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Combined Categories - Frequencies
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). Scores were combined to provide number of participants who indicated they were "worse" (scores of 5, 6, or 7), "no change" (score of 4), or "better" (scores of 1, 2, or 3).
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 48 | 49 | 48
participants
  Worse | 1 | 1 | 3
  No Change | 10 | 5 | 7
  Better | 37 | 43 | 38
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.176, Cochran-Mantel-Haenszel — P-value based on Cochran-Mantel-Haenszel Test with modified ridit scores controlling for alpha block use (yes/no) and lower urinary tract symptom severity as stratification factors
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.921, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]

8. Secondary Outcome: Clinician Global Impression of Improvement (CGI-I) Combined Categories - Frequencies
Description: Measures clinician's perception of patient improvement of illness at the time of assessment compared with start of treatment. Scores range from 1 (very much better) to 7 (very much worse). Scores were combined to provide number of participants whose clinician indicated they were "worse" (scores of 5, 6, or 7), "no change" (score of 4), or "better" (scores of 1, 2, or 3).
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 48 | 49 | 48
participants
  Worse | 0 | 0 | 4
  No Change | 5 | 8 | 4
  Better | 43 | 41 | 40
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.429, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.304, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]

9. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Total, Waking, and Sleeping Voids (Average Number Per Week) Based on Median as Reported in Patient Voiding Dribble Diary
Description: Patient-completed diary that measures daytime frequency (waking voids) and nocturia (sleeping voids). Average number of waking voids per week, average number of sleeping voids per week, and average number of total voids (sleeping+waking) per week are reported.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: average number per week
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 50 | 50 | 49
average number per week
  Baseline Waking Voids | 48.2 (11.2) | 46.9 (11.1) | 48.4 (16.9)
  12 Week Change Waking Voids | -0.3 (8.7) | -2.1 (8.7) | -1.3 (7.6)
  Baseline Sleeping Voids | 10.3 (7.8) | 9.8 (6.7) | 7.9 (5.4)
  12 Week Change Sleeping Voids | -1.3 (3.5) | -2.3 (3.8) | -1.4 (4.0)
  Baseline Total Voids | 58.6 (13.0) | 56.7 (13.3) | 56.3 (19.2)
  12 Week Change Total Voids | -1.6 (9.2) | -4.4 (9.7) | -2.7 (8.9)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.254, Wilcoxon Rank Sum — P-value for 12 Week Change Waking Voids. Change=Endpoint minus baseline. P-values for pairwise comparison of change difference based on Wilcoxon Rank Sum test
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.359, Wilcoxon Rank Sum — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.098, Wilcoxon Rank Sum — P-value for 12 Week Change Sleeping Voids. Change=Endpoint minus baseline. P-values for pairwise comparison of change difference based on Wilcoxon Rank Sum test
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.632, Wilcoxon Rank Sum — [p-value comment as in outcome 9, analysis 3]
Statistical Analysis 5: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.102, Wilcoxon Rank Sum — P-value for 12 Week Change Total Voids. Change=Endpoint minus baseline. P-values for pairwise comparison of change difference based on Wilcoxon Rank Sum test
Statistical Analysis 6: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.348, Wilcoxon Rank Sum — [p-value comment as in outcome 9, analysis 5]

10. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Total Urinary Incontinence Episodes Per Week Based on Median as Reported in Patient Voiding Dribble Diary
Description: A patient-completed diary that measures urinary incontinence (UI) (leaks). Number of UI leaks per week are reported.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: average number per week
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 50 | 50 | 49
average number per week
  Baseline | 0.8 (3.6) | 1.1 (5.4) | 1.6 (5.0)
  12 Week Change | -0.3 (3.5) | 0.7 (2.5) | -0.3 (4.9)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.208, Wilcoxon Rank Sum — P-value for 12 Week Change. Change=Endpoint minus baseline. P-values for pairwise comparison of change difference based on Wilcoxon Rank Sum test
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.985, Wilcoxon Rank Sum — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Voids With Terminal Micturition Dribble and Post Micturition Dribble Per Week Based on Median as Reported by Patient Voiding Dribble Diary
Description: A patient-completed diary that measures terminal dribble (dribble in the end of urination) and post-micturition dribble (dribble after urination).
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: average number per week
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 50 | 50 | 49
average number per week
  Baseline Terminal Micturation Dribble | 68.7 (35.8) | 69.8 (37.0) | 77.5 (29.9)
  12 Week Change Terminal Micturation Dribble | -11.7 (36.9) | 1.6 (31.9) | -8.5 (33.1)
  Baseline Post Micturation Dribble | 14.3 (27.0) | 17.8 (29.8) | 25.5 (32.6)
  12 Week Change Post Micturation Dribble | -0.8 (29.5) | -4.8 (27.4) | -7.6 (34.9)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.385, Wilcoxon Rank Sum — P-value for 12 Week Change Terminal Micturation Dribble. Change=Endpoint minus baseline. P-values for pairwise comparison of change difference based on Wilcoxon Rank Sum test
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.595, Wilcoxon Rank Sum — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.704, Wilcoxon Rank Sum — P-value for 12 Week Change Post Micturation Dribble. Change=Endpoint minus baseline. P-values for pairwise comparison of change difference based on Wilcoxon Rank Sum test
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.439, Wilcoxon Rank Sum — [p-value comment as in outcome 11, analysis 3]

12. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Uroflowmetry Parameters - Peak Urine Flow Rate (Qmax) and Mean Urine Flow Rate (Qmean)
Description: Qmax: defined as the peak urine flow rate (measured in milliliters per second [mL/second] using a standard calibrated flowmeter); and Qmean, defined as the mean urine flow rate (measured in mL/second using a standard calibrated flowmeter).
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliters per second
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 48 | 49 | 48
milliliters per second
  Baseline Qmax | 10.5 (3.6) | 11.4 (3.2) | 11.7 (4.6)
  12 Week Change Qmax | 2.8 (5.6) | 2.4 (5.2) | 1.9 (4.8)
  Baseline Qmean | 5.7 (2.3) | 6.1 (2.1) | 6.2 (3.0)
  12 Week Change Qmean | 2.0 (3.1) | 1.5 (2.9) | 1.0 (3.4)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.838, ANCOVA — P-value for 12 Week Change Qmax. Change=Endpoint minus baseline. P-values are from an ANCOVA with effects for treatment, prior alpha blocker use (yes/no), and baseline value, and were not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.831, ANCOVA — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.696, ANCOVA — P-value for 12 Week Change Qmean. Change=Endpoint minus baseline. P-values are from an ANCOVA with effects for treatment, prior alpha blocker use (yes/no), and baseline value, and were not adjusted for multiple comparisons
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.257, ANCOVA — [p-value comment as in outcome 12, analysis 3]

13. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Uroflowmetry Parameters - Voided Urine Volume (Vcomp)
Description: Vcomp, defined as the volume of voided urine (measured in milliliters [mL]).
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo | Tadalafil | Tamsulosin
Number analyzed (Participants) | 48 | 49 | 48
milliliters
  Baseline | 220.0 (67.7) | 233.2 (86.7) | 236.6 (78.4)
  12 Week Change | 21.4 (128.9) | 19.7 (109.2) | 23.9 (89.3)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.709, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin; Test type: Superiority or Other; p = 0.494, ANCOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Placebo | Tadalafil | Tamsulosin
Serious Adverse Events (participants affected / at risk) | 0 | 2 | 2
Other Adverse Events (participants affected / at risk) | 2 | 4 | 11
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Tadalafil | Tamsulosin
Acute myocardial infarction (Cardiac disorders) | 0/51 (0) | 0/51 (0) | 1/49 (1)
Inguinal hernia (Gastrointestinal disorders) | 0/51 (0) | 0/51 (0) | 1/49 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0/51 (0) | 1/51 (1) | 0/49 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/51 (0) | 1/51 (1) | 0/49 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/51 (0) | 1/51 (1) | 0/49 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Tadalafil | Tamsulosin
Dyspepsia (Gastrointestinal disorders) | 0/51 (0) | 0/51 (0) | 1/49 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0/51 (0) | 0/51 (0) | 1/49 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0/51 (0) | 0/51 (0) | 1/49 (1)
Chest pain (General disorders) | 0/51 (0) | 0/51 (0) | 1/49 (1)
Nasopharyngitis (Infections and infestations) | 0/51 (0) | 1/51 (1) | 5/49 (5)
Intentional overdose (Injury, poisoning and procedural complications) | 0/51 (0) | 1/51 (1) | 1/49 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0/51 (0) | 0/51 (0) | 1/49 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0/51 (0) | 0/51 (0) | 1/49 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/51 (0) | 0/51 (0) | 1/49 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/51 (0) | 2/51 (2) | 1/49 (1)
Headache (Nervous system disorders) | 1/51 (1) | 0/51 (0) | 0/49 (0)
Insomnia (Psychiatric disorders) | 1/51 (1) | 0/51 (0) | 0/49 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0/51 (0) | 1/51 (1) | 0/49 (0)
Flushing (Vascular disorders) | 0/51 (0) | 1/51 (1) | 0/49 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days